CLINICAL TRIAL: NCT00767182
Title: Estimation of the Placental Volume by 3D Ultrasound at 12, 16 and 22 Weeks : Relation With Growth Factors and D-Dimers - Monocentric Prospective Cohort
Brief Title: Estimation of the Placental Volume by 3D Ultrasound at 12, 16 and 22 Weeks : Relation With Growth Factors and D-Dimers
Acronym: VOLUPLA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Groupe de Recherche sur la Thrombose (Other)
Responsible Party: Sponsor
Other Study IDs: 0808025; 2008-A00233-52 (Other: ANSM); DGS2008-0193 (Other: DGOS)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Placenta Vascular Malformation
Keywords: preeclampsia; eclampsia; retroplacental hematoma; vascular IUGR; IUFD; placental volume
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant patients with VPP antecedent: Pregnancy women consulting for an scan during their 12th week of amenorrhea at the University Hospital of Saint Etienne will be studied in this clinical trial. They have an history of VPP (Vascular Placental Pathology). They will have to give a blood sample.
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — biological markers evaluated : D-Dimer, sEPCR

SUMMARY:
Pregnancy complications called PVP are mainly responsible for perinatal mortality. In these cases, the placenta is smaller and often the centre of thrombotic lesions. The estimation of the placenta volume by 3D ultrasound coupled with growth factors and D-Dimers measures could improve the understanding of these pathologies to optimize their detection.

DETAILED DESCRIPTION:
Pregnancy complications called Placental Vascular Pathologies (PVP) are mainly responsible for perinatal mortality. In these cases, the placenta is smaller and often the centre of thrombotic lesions. The estimation of the placenta volume by 3D ultrasound coupled with growth factors and D-Dimers measures could improve the understanding of these pathologies to optimize their detection. Thus, the identification of predictive factors of the risk of occurrence or recurrence of PVP could allow us to propose a monitoring of patients at risk, to anticipate corticoids administration for the foetuses pulmonary maturation and perhaps later to adapt anti hypertensive and antithrombotic therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* previous history of one or more PVC episodes : preeclampsia, HELLPs, retroplacental hematoma, vascular IUGR<10th percentile, recurrence miscarriage >2, unexplained IUFD or IUFD after abruption placentae, eclampsia.
* coming for a 12 weeks ultrasound

Exclusion Criteria:

* Multiple pregnancy
* past history of in utero fetal death due to congenital malformations, rhesus incompatibility or an infection
* previous history of IUGR which etiology was a chromosomal, genic or infectious anomaly

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
placental volume by 3D ultrasound and D-Dimers rate | Week 12

SECONDARY OUTCOMES:
EPCRs rate measurements | Week 12
EPCRs rate measurements | Week 16
EPCRs rate measurements | Week 22
Occurrence or recurrence of PVP | Week 12
Occurrence or recurrence of PVP | Week 16
Occurrence or recurrence of PVP | Week 22
placental volume by 3D ultrasound and D-Dimers rate | Week 16
placental volume by 3D ultrasound and D-Dimers rate | Week 22

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Service de Gynécologie Obstétrique - CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No